CLINICAL TRIAL: NCT02571335
Title: Intensity-dependent Impacts of Training on Growth Factors BDNF and Cognitive Functions in Persons With Multiple Sclerosis - a Single-center Randomized Controlled Trial
Brief Title: Impacts of Different Training Modes (Intense Versus Ordinary) on the Immune System and Memory Functions in pwMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik Valens (Other)
Collaborators: German Sport University, Cologne (Other)
Responsible Party: Principal Investigator, Jens Bansi, Exercise Sciences, PhD, Klinik Valens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: JBansi
Record Dates: First submitted 2015-09-23; First posted 2015-10-08 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Training (Experimental): Treatment consists of endurance training in both groups of physiologically defined heart rate controlled cycling at 50-60 rounds per minutes (rpm) and progressive resistance training. Training groups differ in the applied intensities and frequencies.The IT will train less frequent but training sessions will be more intensive in its effects. Training will be performed daily in six sessions (three morning and three afternoon sessions), synchronized and individually matched to a ratio of active versus passive sessions of 2:1.
  Interventions: Behavioral: Intensive Training
- Normal Training (Active Comparator): The NT is the normal training performed out of the daily routine and outlines the usual care of the Valens clinic. Training will be performed in up to eight training sessions that will not be synchronized and not individually matched to a ratio of active versus passive sessions.
  Interventions: Behavioral: Normal Training

INTERVENTIONS:
Behavioral: Intensive Training — Week 1: Ratio of continuous and interval training of 2:1. Entry point at day one with 20 min of continuous, physiologically defined heart rate controlled cycling at 50-60 rounds per minutes at 75% of HRpeak.
  Resistance training is performed with 70% of the subjective-felt 1-round maximum with three sets and 10-12 repetitions and three exercises for the upper and lower extremities.
  Week 2 Progression of endurance training: 4x5 minutes with 2 Minutes between each interval performed at 80% of HRmax Progression resistance training: 75% of the subjective-felt 1-round maximum with three sets and 8-10 repetitions and three exercises for the upper and lower extremities.
  Week 3 Same as week 2.
  Other Names: Endurance and Resistance Training
  Arms: Intensive Training
Behavioral: Normal Training — The control intervention is the normal rehabilitation program of the Valens clinic.
  Other Names: Endurance and Resistance Training
  Arms: Normal Training

SUMMARY:
Multiple Sclerosis (MS) is a chronic immune-mediated disease of the central nervous system, accompanied by varying inflammatory manifestations, demyelinization and axonal loss. With chronic progressive or relapsing-remitting disease onsets persons with MS (pwMS) progressively develop impaired functional capacity and show reduced physical activity and cognitive decline compared to healthy controls. The primary aims of rehabilitation in pwMS are therefore to increase levels of activity and participation leading to increase independence of the participants. In general exercise ranges from passive physiotherapy-based interventions to submaximal endurance training sessions. Current recommendations advise pwMS that exercise should be matched with the individual performance capacities. Exercise training in pwMS then has the potential to target and improve many components outlined in the ICF-model.

Cytokines and neurotrophic factors have received increased attention in MS research and addressed the brain-derived neurotrophic factor (BDNF) as an important mediator of neuronal regeneration linking the effects of exercise with MS pathogenesis. Data show positive connections between elevated neurotrophin concentrations, induction of neuroplasticity, recovery of the motor and cognitive functions and the applied training intensities. Similarly, intensive and progressive exercise bouts seem to have greater benefits on cardiorespiratory fitness and maximum voluntary strength in elderly and seniors with dementia. Therefore, specific exercise prescriptions may be necessary for targeting the specific impairments also in pwMS.

This study aims to evaluate two different training modalities (intensive versus normal) in pwMS. It is expected that both modalities will improve cardiorespiratory fitness and cognitive functions in pwMS. Based on the findings that higher training intensities facilitate greater benefits, it is expected that pwMS will tolerate the intensive training intensities and show positive connections to elevated neurotrophin concentrations.

The results will to help to clearer understand the benefits of each type of exercise conveyed for pwMS and will assist in the development of patient-specific exercise prescriptions.

DETAILED DESCRIPTION:
This study aims to evaluate two different training modalities (intensive versus normal) in pwMS. It is expected that both modalities will improve cardiorespiratory fitness and cognitive functions in pwMS. Based on the findings that higher training intensities facilitate greater benefits, it is expected that pwMS will tolerate the intensive training intensities and show positive connections to elevated neurotrophin concentrations.

Primary outcomes are the acute (after CPET) and chronic (3-week training intervention) changes of neurotrophic factors and cognitive functions. All other measures are secondary outcomes (Training values: VO2peak, Workload, Heart rate; Fatigue: FSMC; Anxiety and Depression: HADS.

Participants are eligible if they hold a definite diagnosis of multiple sclerosis (revised McDonald criteria), an EDSS score of 1.0 -6.0, they give no written consent, severe cardiovascular exacerbations (RR > 240/120, HR above the age predicted maximum of 220-Age) are persistent, they hold severe cognitive impairments, they face severe disease progression or relapses.

Main measurements and procedures include:

Blood sampling: Blood samples (10ml) of the primary outcomes will be taken by vein puncture from the antecubital vein in a seated position before the exercise bout and straight after reaching VO2peak during cool down, with the participant still seated on the ergometer.

Before samples are taken the participant will be required to relax for 10 minutes, blood sampling will take approximately 5 minutes.

Cardiopulmonary Exercise Test (CPET): Cardiorespiratory fitness is assessed through a progressive CPET performed at baseline on a cycle ergometer at t1 and is repeated the day prior to discharge at t2.

The exercise protocol consists of (a) first 3 minutes at rest (no pedalling) on the cycle ergometer; (b) 3 minutes of unloaded pedalling as a warm up; (c) testing phase until the participant reaches a symptom limited maximum. Workload is continuously ramp type increased by 5-10 Watts every minute to ensure 8-12 minutes of testing; (d) the final 3 minutes are unloaded pedalling to cool down. Heart rate (Polar Electro, Kempele, Finland) and blood pressure (Riva-Rocci) are monitored for the last 10 seconds every 2 minutes during the test. The 10-point BORG scale therapy short-form assesses the rate of perceived exertion (RPE) at phases (c) and (d). Blood samples are drawn at rest prior to phase (a) and at the end of CPET phase (d) at t1 and t2

Cognitive assessments: Cognitive assessments will be performed using the German version of the Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS). Additionally, the German version of the Trail-Making-Pencil-Test versions A/B (TMT-A/B) and Go/noGo (TAP version) will be used. Cognitive assessments will be performed at baseline (t1) and repeated at t2.

Fatigue: Fatigue is assessed with the multidimensional FSMC scale before CPET under resting conditions. FSMC has defined cut-off scores to classify mildly, moderately and severely fatigued patients. Cut-off for fatigue is set for the total score at 43 and for the motoric and cognitive sub-scores at 22. The scale has a proven test-retest liability and has been translated into multiple languages.

Depression and Anxiety: Depression and anxiety are assessed with the Hospital Anxiety and Depression Scale (HADS). The HADS is a self-assessment questionnaire for adults with physical ailments that assess anxiety and depression. The questionnaire consists of 14 items seven for anxiety seven for depression with higher scores indicating anxiety or depression.

Training: Endurance training in both groups consisted of physiologically defined heart rate controlled cycling at 50-60 rounds per minutes (rpm) and progressive resistance training. All participants will be stratified according to their cardiorespiratory fitness and level of cognitive fatigue in to group Intensive Training (IT) and Normal Training (NT). Training groups differ in the applied intensities and frequencies.

The IT will train less frequent but training sessions will be more intensive in its effects. Training will be performed daily in six sessions (three morning and three afternoon sessions), synchronized and individually matched to a ratio of active versus passive sessions of 2:1.

The NT is the normal training performed out of the daily routine and outlines the usual care of the Valens clinic. Training will be performed in maximal eight training sessions and will not be synchronized and not individually matched to a ratio of active versus passive sessions.

ELIGIBILITY:
Inclusion Criteria:

Key inclusion criteria for the participants' eligibility are a definite MS diagnosis (McDonald criteria). Participants fulfilling the key inclusion and the following criteria are eligible for this study

* EDSS 1.0 - 6.0
* Age 19 - 75 years

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* Persistent infections
* Severe cardiovascular and pulmonal diseases (renal failure, hepatic dysfunction, cardiovascular disease)
* Severe cardiovascular exacerbations (RR > 240/120, HR above the age predicted maximum of 220-Age) during training
* Immunosuppressive therapy the day of CPET
* Life style factors and / or persistent addictions (drug or alcohol abuse)
* Inability to follow the study procedures (due to psychological disorders or dementia)
* Insufficient knowledge of the project language (German)
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his / her family members, employees and other dependent persons,
* Specific exclusions for the disease under study,
* Specific concomitant therapy washout requirements prior to and/or during study participation,
* Dietary restrictions

Exclusion Criteria: Criteria in which the participant withdraws from this study may be the following:

* Inability to comply with the daily schedule
* Strong symptom exacerbations
* Withdrawal of informed consent
* Non-compliance
* Disease progression or relapse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Neurotrophic Factor BDNF | 3-weeks
  Short- and long-term changes (pg/ml) of serum levels of the neurotrophic factor BDNF (t1-->t2)

SECONDARY OUTCOMES:
Maximum Oxygen consumption (VO2peak) | 3-weeks
  workload (W) achieved in the cardiopulmonary exercise test.
Maximum heart rate (HRmax) | 3-weeks
  Changes in beats min-1 over three weeks training
Maximum workload (Loadmax) | 3-weeks
  Changes in Watt over three weeks training
Fatigue | 3-weeks
  Changes over three weeks Training of Motor and Cognitive fatigue (Cut-off for fatigue is set for the total score at 43 and for the motoric and cognitive subscores at 22).
Health-related Quality of life | 3-weeks
  Changes of anxiety and Depression over three weeks Training (Cut off for anxiety and Depression are set at 4 Points
Cognitive Functions | 3-weeks
  Cognitive functions will be the changes on the Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) and the Trail-Making-Pencil-Test versions A/B (TMT-A/B) both performed at baseline (t1) and repeated at t2

CONTACTS AND LOCATIONS:
Overall Officials: Juerg Kesselring, Prof, Study Chair — Klinik Valens
Locations (1):
- Kliniken-Valens, Valens, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zimmer P, Bloch W, Schenk A, Oberste M, Riedel S, Kool J, Langdon D, Dalgas U, Kesselring J, Bansi J. High-intensity interval exercise improves cognitive performance and reduces matrix metalloproteinases-2 serum levels in persons with multiple sclerosis: A randomized controlled trial. Mult Scler. 2018 Oct;24(12):1635-1644. doi: 10.1177/1352458517728342. Epub 2017 Aug 21. PMID 28825348